CLINICAL TRIAL: NCT02343380
Title: Is the Timing of Caloric Intake Associated With Variation in Diet-induced Thermogenesis and Hormonal Pattern?
Brief Title: Timing of Caloric Intake, Diet-induced Thermogenesis and Hormonal Pattern
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Simona Bo, Professor Assistant, MD, University of Turin, Italy
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: DIT-01
Record Dates: First submitted 2015-01-12; First posted 2015-01-22 (Estimated); Results first posted 2015-12-31 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Diet-induced Thermogenesis
Keywords: diet-induced thermogenesis; glucose; respiratory quotient

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- morning-first (Experimental): calorimetric exam after a standard meal
  Interventions: Other: calorimetric exam after a standard meal
- evening-first (Experimental): calorimetric exam after a standard meal
  Interventions: Other: calorimetric exam after a standard meal

INTERVENTIONS:
Other: calorimetric exam after a standard meal — The calorimetric and metabolic responses to identical meals (a high-protein, low-carbohydrates meal) consumed in the morning (8:00 am) and in the evening (8:00 pm) are measured in healthy volunteers, after standardizing diet, physical activity level, duration of fast and resting

SUMMARY:
The investigators aim at analyzing whether eating a standard meal in the evening (at 8:00 pm) determines in the same individuals a lower diet-induced thermogenesis (DIT) and a different hormonal response than the consumption of the same meal in the morning (at 8:00 am).

The primary outcome is: the intra-individual variation in DIT after the evening and morning meal consumption.

The secondary outcomes are the intra-individual variations in glucose, triglyceride, insulin, free fatty acids, leptin, glucagon-like peptide-1, acylated ghrelin, adrenalin, noradrenalin, after the evening and morning meal consumption.

DETAILED DESCRIPTION:
Twenty healthy volunteers (ten males and ten females) are recruited among students and graduates attending the Department of Medical Sciences of Turin (Italy) to take part to this randomized cross-over trial.

Participants randomly receive first the standard meal at 8:00 am and the week after the standard meal at 8:00 pm or vice versa. Eight-h before the meal (respectively at 12:00 pm or at 12:00 am), the participants receive the same standard meal (without protein supplementation) at their home, and then are asked to spend in bed the following 6 hours. A 24-h urine collection is collected the day before each test in order to determine total urinary nitrogen excretion.

The standard meal consists of: 100g white bread, 100g ham, 50g cheese, 125g yogurt, 200ml fruit juice, plus 25g protein supplement. The participants must consume each meal in 25-30 minutes.

A 30-min basal calorimetric (Deltatrac II) exam is performed. Participants remain in a supine position but awake and motionless on a hospital bed during the whole period, except during the meal, when they can sit to eat. At 8:00 am (or pm), the participants consume the meal, and then rest in a supine position for 90 min. Then, a second 60 min-calorimetric evaluation is done. From the first calorimetric exam (the basal) until the end of the second (post-prandial) blood samples are drawn every 30 min. The same time schedule is adopted in the case of the morning meal (at 8:00 am) and the evening meal (at 8:00 pm).

The random sequence (morning/evening, evening/morning meal) is computer-generated, using blocks of different lengths in random order.

The following are measured: weight, height, waist circumference, and at baseline and every 30-min during the morning and evening tests: glucose, triglyceride, insulin, free-fatty acids, leptin, glucagon-like peptide-1, acylated ghrelin, adrenalin, noradrenalin.

ELIGIBILITY:
Inclusion Criteria:

* body mass index 19-26 kg/m2
* habitual moderate exercise level

Exclusion Criteria:

* any acute or chronic diseases
* menopause
* any drugs or supplementations
* any alimentary restrictions or specific diets
* being a shift or night workers
* unable to give a written informed consent

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-05; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simona Bo, MD, Principal Investigator — University of Turin, Italy

REFERENCES:
- [Derived] Bo S, Fadda M, Castiglione A, Ciccone G, De Francesco A, Fedele D, Guggino A, Parasiliti Caprino M, Ferrara S, Vezio Boggio M, Mengozzi G, Ghigo E, Maccario M, Broglio F. Is the timing of caloric intake associated with variation in diet-induced thermogenesis and in the metabolic pattern? A randomized cross-over study. Int J Obes (Lond). 2015 Dec;39(12):1689-95. doi: 10.1038/ijo.2015.138. Epub 2015 Jul 29. PMID 26219416

RESULTS

PARTICIPANT FLOW:
Groups:
- Morning-first, Then Evening; Evening-first, Then Morning: calorimetric exam after a standard meal
  calorimetric exam after a standard meal: The calorimetric and metabolic responses to identical meals (a high-protein, low-carbohydrates meal) consumed in the morning (8:00 am) and in the evening (8:00 pm) are measured in healthy volunteers, after standardizing diet, physical activity level, duration of fast and resting
Period: Overall Study
Arm/Group | Morning-first, Then Evening | Evening-first, Then Morning
Started | 10 (Morning test (first week)) | 10 (Evening test (first week))
Completed | 10 (Evening test (second week)) | 10 (Morning test (second week))
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Morning-first, Then Evening | Evening-first, Then Morning | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.9 (3.3) | 27.4 (3.6) | 27.6 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 5 | 5 | 10
fasting Resting Metabolic rate [Mean (Standard Deviation); unit: Kcal/min] | 1545.0 (266.8) | 1540.0 (235.0) | 1543.5 (244.7)

OUTCOME MEASURES:

1. Primary Outcome: Intra-individual Variation in Morning Diet-induced Thermogenesis (DIT) Evaluated by Calorimetric Exam After the Consumption of a Meal at 8:00 am Compared With Evening DIT Evaluated by Calorimetric Exam After the Consumption of the Same Meal at 8:00 pm
Description: Indirect calorimetry by Deltatrac II (DATEX, Division of Instruments Corp. Helsinki, Finland) is used to measure the rate of energy expenditure before- and after- the meal.Diet-induced thermogenesis is considered as the difference between average after-meal and basal energy expenditure.
Time Frame: Before and 180-min from the beginning of the meal
Measure: Mean (95% Confidence Interval); unit: kcal/min
Groups:
- Morning; Evening: calorimetric exam after a standard meal
  calorimetric exam after a standard meal: The calorimetric and metabolic responses to identical meals (a high-protein, low-carbohydrates meal) consumed in the morning (8:00 am) and in the evening (8:00 pm) are measured in healthy volunteers, after standardizing diet, physical activity level, duration of fast and resting
Arm/Group | Morning | Evening
Number analyzed (Participants) | 20 | 20
kcal/min | 327.5 [279.0 to 376.0] | 237.0 [195.1 to 278.9]

2. Secondary Outcome: Variation in Morning Glucose and Insulin Area-Under the Curve (AUC)s After the Consumption of a Meal at 8:00 am Compared With Evening Glucose and Insulin AUCs After the Consumption of the Same Meal at 8:00 pm
Description: Glucose and insulin values measured every 30 minutes after meal for 180-min. Time 0 was before the meal. Times 30, 60, 90, 120, 150 and 180 were referred to the time intervals in minutes from the beginning of the meal. AUCs were calculated according to the trapezoidal model.
  Serum glucose was measured by enzymatic colorimetric assay; serum insulin was determined by immunoradiometric assay.
Time Frame: From the beginning of the meal for 180-min
Measure: Mean (95% Confidence Interval); unit: ug/ml*h
Groups:
- Morning: Variation in morning glucose and insulin Area-Under the Curve (AUC)s after the consumption of a meal at 8:00
- Evening: Variation in morning glucose and insulin Area-Under the Curve (AUC)s after the consumption of a meal at 8:00 pm
Arm/Group | Morning | Evening
Number analyzed (Participants) | 20 | 20
ug/ml*h
  Glucose AUCs | 15383 [14426 to 16340] | 17183 [16111 to 18255]
  Insulin AUCs | 6969 [5664 to 8274] | 8598 [6618 to 10578]

3. Secondary Outcome: Variation in Morning Triglyceride and Free Fatty Acid (FFA) Area-Under the Curve (AUC)s After the Consumption of a Meal at 8:00 am Compared With Evening Glucose and Insulin AUCs After the Consumption of the Same Meal at 8:00 pm
Description: Triglycerides and FFA values measured every 30 minutes after meal for 180-min. Time 0 was before the meal. Times 30, 60, 90, 120, 150 and 180 were referred to the time intervals in minutes from the beginning of the meal. AUCs were calculated according to the trapezoidal model.
  FFA concentrations were measured by a fluorometric assay. Plasma triglycerides were assayed by enzymatic colorimetric method.
  Serum glucose was measured by enzymatic colorimetric assay; serum insulin was determined by immunoradiometric assay.
Time Frame: From the beginning of the meal for 180-min
Measure: Mean (95% Confidence Interval); unit: mmol/l*h
Groups:
- Morning: Variation in morning triglyceride and free fatty acid (FFA) Area-Under the Curve (AUC)s after the consumption of a meal at 8:00 am.
  The metabolic responses to identical meals (a high-protein, low-carbohydrates meal) consumed in the morning (8:00 am) and in the evening (8:00 pm) are measured in healthy volunteers, after standardizing diet, physical activity level, duration of fast and resting
- Evening: Variation in morning triglyceride and free fatty acid (FFA) Area-Under the Curve (AUC)s after the consumption of a meal at 8:00 pm
  The metabolic responses to identical meals (a high-protein, low-carbohydrates meal) consumed in the morning (8:00 am) and in the evening (8:00 pm) are measured in healthy volunteers, after standardizing diet, physical activity level, duration of fast and resting
Arm/Group | Morning | Evening
Number analyzed (Participants) | 20 | 20
mmol/l*h
  triglyceride AUCs | 11721 [9794 to 13648] | 12363 [11068 to 13658]
  FFA AUCs | 38.7 [30.9 to 46.5] | 54.7 [40.6 to 68.9]

4. Secondary Outcome: Intra-individual Variations in the Values of Adrenalin and Noradrenalin, After the Morning and Evening Meal Consumption
Time Frame: Every 30-min from the beginning of the meal for 180-min
Measure: Mean (95% Confidence Interval); unit: ng/l x h
Groups:
- Morning: Variation in morning adrenalin and noradrenalin Area-Under the Curve (AUC)s after the consumption of a meal at 8:00 am
- Evening: Variation in evening adrenalin and noradrenalin Area-Under the Curve (AUC)s after the consumption of a meal at 8:00
Arm/Group | Morning | Evening
Number analyzed (Participants) | 20 | 20
ng/l x h
  adrenalin | 4543.5 [3204.6 to 5882.4] | 3020.7 [2618.4 to 3423.0]
  noradrenalin | 37504.9 [32516.8 to 42492.9] | 32718.4 [25987.6 to 39449.3]

5. Secondary Outcome: Intra-individual Variations in the Values of Acylated Ghrelin After the Morning and Evening Meal Consumption
Time Frame: Every 30-min from the beginning of the meal for 180-min
Measure: Mean (95% Confidence Interval); unit: ng/l x h
Groups:
- Morning: Variation in morning acylated ghrelin Area-Under the Curve (AUC)s after the consumption of a meal at 8:00 am
- Evening: Variation in evening acylated ghrelin Area-Under the Curve (AUC)s after the consumption of a meal at 8:00 pm
Arm/Group | Morning | Evening
Number analyzed (Participants) | 20 | 20
ng/l x h | 8013.5 [6190.4 to 9836.7] | 9631.3 [7296 to 11966.6]

6. Secondary Outcome: Intra-individual Variations in the Values of Glucagon-like Peptide-1 After the Morning and Evening Meal Consumption
Time Frame: Every 30-min from the beginning of the meal for 180-min
Population: These variables were not measured, since data were not collected.
Groups:
- Morning: Variation in morning glucagon-like peptide 1 Area-Under the Curve (AUC)s after the consumption of a meal at 8:00 am
- Evening: Variation in morning glucagon-like peptide 1 Area-Under the Curve (AUC)s after the consumption of a meal at 8:00
Arm/Group | Morning | Evening
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: The day of each test
Arm/Group | Morning | Evening
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No